CLINICAL TRIAL: NCT02775123
Title: Cytokine Clearance With Cytoabsorbant Device During Cardiac Bypass: a Pilot Study
Brief Title: Cytokine Clearance With Cytoabsorbant Device During Cardiac Bypass
Acronym: CCCC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Antoine Schneider, physician associate, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2015-00010
Record Dates: First submitted 2016-04-21; First posted 2016-05-17 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Myocardial Ischemia; Heart Valve Diseases
MeSH Terms: conditions — Myocardial Ischemia; Heart Valve Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Conventional cardio-pulmonary bypass
- Cytosorb (Experimental): Cytosorb added to cardio-pulmonary bypass
  Interventions: Device: Cytosorb

INTERVENTIONS:
Device: Cytosorb — A cytoadsorbent cardridge (Cytosorb) will be added to the extra-corporeal circuit (CPB).
  Arms: Cytosorb

SUMMARY:
Investigators are planning a single center pilot randomized controlled trial to assess the potential of a Cytoadsorbant filter (Cytosorb®, Germany) to remove cytokines from the blood during cardiac surgery.

Investigators will screen all patients undergoing cardiac surgery and approach those deemed at risk of post surgical complications [≥ 1 among: age >75 years old, double valvular replacement, complex surgery with expected CPB time >100 min, redo cardiac surgery, pre-op chronic renal failure (plasma creatinine level >120 mcmol/l) or chronic heart failure (LVEF <35%)].

Patients with end-stage renal disease (dialysis dependence), undergoing an emergency procedure or an off-pump procedure, those who decline informed consent as well as those enrolled in another conflicting study will be excluded.

Eligible patients will be approached, consented and enrolled in the trial. Patients will then be randomized to either receive conventional CPB (control arm) or CPB plus Cytosorb (intervention arm). The target population is 30 patients (15 per arm).

For this pilot study, investigators main outcome will be differences between the two arms in measurement of serum levels for IL-2, IL-6, IL-10 and TNF alpha at baseline (pre-operatively), on ICU admission, as well as 6 and 24 hrs post CPB.

Secondary outcomes will be changes in coagulation factors serum levels, the need for vasopressors, inotropes, mechanical ventilation and renal replacement therapy, ICU and hospital length of stay as well as in-hospital mortality.

Recruitment period should span from May 2016 to April 2017.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned for elective cardiac surgery requiring CPB and (≥1 among):

  * Age >75 years' old AND / OR
  * Double valvular replacement AND / OR
  * Complex surgery with expected CPB time >120 min AND / OR
  * Redo cardiac surgery AND / OR
  * Pre-op chronic renal failure (GFR<30 ml/min) AND / OR Chronic heart failure (LVEF <40%)

Exclusion Criteria:

* End stage renal disease (dialysis dependence)
* Emergency procedure
* Active infectious endocarditis
* Off-pump procedure planned
* Non steroidal anti-inflammatory treatment in the previous 7 days
* Corticosteroids administration in the previous 7 days
* No informed consent
* Enrolment in another conflicting study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Change in Cytokine levels | From Baseline (Preoeratively) to 6hrs post CPB

SECONDARY OUTCOMES:
Change in Cytokine levels | From Baseline (Preoeratively) to 24 hrs post CPB
Change in Cytokine levels | From Baseline (Preoeratively) to end of CPB
Change in Coagulation factors serum levels | From baseline (pre-operatively) to end of CPB as well as 6 hrs and 24 hrs post CPB
Duration of the need for vasopressors | 28 days
Duration of mechanical ventilation | 28 days
ICU length of stay | 90 days
Hospital Length of stay | 90 days
In-hospital mortality | 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Poli EC, Alberio L, Bauer-Doerries A, Marcucci C, Roumy A, Kirsch M, De Stefano E, Liaudet L, Schneider AG. Cytokine clearance with CytoSorb(R) during cardiac surgery: a pilot randomized controlled trial. Crit Care. 2019 Apr 3;23(1):108. doi: 10.1186/s13054-019-2399-4. PMID 30944029